CLINICAL TRIAL: NCT05127577
Title: Effect of Abdominal Massage on Excretory Activity and Pulmonary Function Tests in Patients With Partial Hip Replacement
Brief Title: Effect of Abdominal Massage on Excretory Activity and Pulmonary Function Tests in Patients After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Canan KANAT, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinUCKANAT-01
Record Dates: First submitted 2021-10-27; First posted 2021-11-19 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Intraabdominal Pressure
Keywords: Abdominal massage; Pulmonary function tests; Partial hip replacement; Nursing care; Excretory activity; Defecation

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm, randomized controlled clinical trial
Who Masked: Participant
Masking Description: According to the randomization table, the information showing the patients included in the research sample is assigned to the A and B groups will be put in an opaque envelope. This envelope will be kept by the coordinator researcher (GAU) and when the researcher (CK) goes to the patient for application, after filling out the "Informed Voluntary Consent Form", he will open the envelope and learn which group is in which group. Due to the nature of the study, patients and the researcher (CK) will not be blinded, since abdominal massage will be applied only to the patients included in the study. When the research is completed, the data will be transferred to the computer environment by a statistician who does not know the A and B groups, and the data will be analyzed by a statistician independent of the research and the findings will be reported. Thus, the data analysis and statistics phase will be blind to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal massage group (Experimental): Abdominal massage will be applied to the experimental group 2 times a day, morning and evening, until defecation, starting in the evening of the first day after the surgical intervention.
  Interventions: Other: Abdominal massage
- Control group (No Intervention): The control group will be received routine treatment and care in the unit.

INTERVENTIONS:
Other: Abdominal massage — Abdominal massage will be applied to patients at least 30 minutes after morning and evening meals (8:30 in the morning, 20:30 in the evening) for 15 minutes each, similar to the literature [33,34,38]. Data of the patients will be collected again 15 minutes after the application of abdominal massage (09:00-09:15 in the morning, 21:00-21:15 in the evening). Abdominal massage will start in the evening of the day the patient is transferred to the clinic (20:30), and will be terminated when the patient defecates. In order to stimulate bowel movements, four basic movements will be used in the abdominal massage to be applied clockwise: superficial effusion, deep effusion, petrissage, and vibration.
  Arms: Abdominal massage group

SUMMARY:
This study is aimed to determine the effect of abdominal massage on excretory activity and pulmonary function tests (PFT) in patients undergoing PKP.

DETAILED DESCRIPTION:
Methods: The research will be carried out with 78 patients who underwent partial hip replacement. Patients were assigned to study (abdominal massage) and control groups by randomization. Abdominal massage will be applied to the patients at least 30 minutes after the morning and evening meals (08:30 in the morning, 20:30 in the evening) for 15 minutes, similar to the literature. Patients' data will be collected 15 minutes before and after the application of abdominal massage. Within the scope of the patient's data, information on pulmonary function test values, intra-abdominal pressure value and excretory activities will be collected. Abdominal massage will start in the evening of the day the patient is transferred to the clinic (20:30), and will be terminated when the patient defecates. No treatment will be applied to the patients in the control group. The data recorded before and after the abdominal massage in the study group will be recorded in the Excretory Activity Form and the Pulmonary Function Test Form as a result of the measurements made at the same time in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Having a urinary catheter for at least one day after surgery,
* Discharged at least 48 hours after surgery,
* Do not have any condition for which abdominal massage is contraindicated (inflammatory bowel disease, presence of abdominal tumor, surgical intervention or radiotherapy to the abdominal region, presence or suspicion of ileus, and pregnancy),
* No diagnosis of chronic constipation made by a physician,
* Who has not developed any respiratory tract complications (atelectasis, pneumonia, etc.) due to surgical intervention,
* No chronic respiratory disease (chronic obstructive pulmonary disease, pulmonary hypertension, sleep apnea syndrome, asthma, chronic bronchitis, cystic fibrosis, occupational lung diseases, etc.),
* Patients who do not have problems in transition to oral feeding and who can be fed orally will be included in the study.

Exclusion Criteria:

* Urinary catheter removed within the first day after surgery,
* Discharged before 48 hours after surgery,
* Any condition in which abdominal massage is contraindicated (inflammatory bowel disease, presence of abdominal tumor, surgical intervention or radiotherapy to the abdominal region, presence or suspicion of ileus, and pregnancy),
* Having a diagnosis of constipation made by a physician,
* Having any respiratory complications (atelectasis, pneumonia, etc.) developed due to surgical intervention,
* Having chronic respiratory disease (chronic obstructive pulmonary disease, pulmonary hypertension, sleep apnea syndrome, asthma, chronic bronchitis, cystic fibrosis, occupational lung diseases, etc.),
* Patients who have problems in the transition to oral feeding and cannot be fed orally will not be included in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Intra-abdominal Pressure Value | up to first defecation an average of 3 days
  Intra-abdominal pressure measurement will be performed using the existing urinary catheter in the patient. This measurement method, which is performed through the bladder, is accepted as the gold standard for intra-abdominal pressure measurement because it is an easy-to-apply and minimally invasive procedure [25,43]. The investigator (CK) will measure the intra-abdominal pressure via a sterile single-transducer pressure monitoring set, which will be attached to the patient's urinary catheter at one end and to a portable monitor capable of measuring pressure at the other end. The measured value will be recorded in Excretory Activities Form.
Return time of bowel sounds | up to first defecation an average of 3 days
  The return time of bowel sounds will be evaluated morning and evening and recorded in the Excretory Activities Form.
Number of bowel sounds | up to first defecation an average of 3 days
  The number of bowel sounds will be evaluated morning and evening and recorded in the Excretory Activities Form.
First defecation time | up to first defecation an average of 3 days
  The time to first defecation will be asked morning and evening after surgery and recorded in the Excretory Activities Form.
Amount of laxative use | up to first defecation an average of 3 days
  The amount of drug use to assist with defecation will be evaluated morning and evening and recorded in the Excretory Activities Form.

SECONDARY OUTCOMES:
Pulmonary Function Tests- FVC | up to first defecation an average of 3 days
  The FVC value obtained using the Respiratory Function Test device will be recorded in the Pulmonary Function Tests Form.
Pulmonary Function Tests- FEV-1 | up to first defecation an average of 3 days
  The FEV-1 value obtained using the Respiratory Function Test device will be recorded in the Pulmonary Function Tests Form.
Pulmonary Function Tests- FEV1/FVC | up to first defecation an average of 3 days
  The FEV1/FVC value obtained using the Respiratory Function Test device will be recorded in the Pulmonary Function Tests Form.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Altun Uğraş, doctorate, Study Director — Mersin University
Locations (1):
- Mersin Univercity, Mersin, Turkey (Türkiye)